CLINICAL TRIAL: NCT03223194
Title: VALENS: A Phase 1/2, Randomized, Open-Label, Ascending-Dose, Delayed-Treatment Concurrent Control Clinical Study to Evaluate the Safety and Preliminary Efficacy of AT342, an AAV8-Delivered Gene Transfer Therapy in Crigler-Najjar Syndrome Subjects Aged 1 Year and Older
Brief Title: Gene Transfer Clinical Study in Crigler-Najjar Syndrome
Acronym: VALENS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Audentes Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AT342-02
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Crigler-Najjar Syndrome
Keywords: Crigler-Najjar; CN; AAV8 Delivered Gene Transfer; Adeno Associated Virus
MeSH Terms: conditions — Crigler-Najjar Syndrome

STUDY DESIGN:
Intervention Model Description: Up to four subjects will be enrolled at each dose level including up to1 subject at each dose level randomized to control with delayed initiation of treatment. One of the dose levels will be chosen for dose expansion and all control subjects will then be treated at the chosen dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 1.5 x 10^12 vg/kg of AT342 delivered intravenously one time
  Interventions: Genetic: AT342
- Cohort 2 (Experimental): 6.0 x 10^12 vg/kg of AT342 delivered intravenously one time
  Interventions: Genetic: AT342
- Cohort 3 (Experimental): 1.5 x 10^13 vg/kg of AT342 delivered intravenously one time
  Interventions: Genetic: AT342
- Delayed-Treatment Control (No Intervention): Control subjects will generally have the same assessments as treated subjects. Once the optimal dose is selected, control subjects will undergo pre-treatment baseline procedures to confirm that they are eligible to receive treatment with AT342. Once eligible control subjects are dosed with AT342, they will initiate the same post-dose procedures as subjects who received AT342.

INTERVENTIONS:
Genetic: AT342 — AT342 is an AAV8 vector containing a functional copy of the UGT1A1 gene.
  Arms: Cohort 1; Cohort 2; Cohort 3

SUMMARY:
This is a Phase 1/2, multinational, open-label, ascending-dose, delayed-treatment concurrent control clinical study to evaluate the safety and preliminary efficacy of AT342 in subjects with Crigler-Najjar aged ≥1 year. Subjects will receive a single dose of AT342 and will be followed for safety and efficacy for 5 years.

DETAILED DESCRIPTION:
This study will evaluate safety and preliminary efficacy of gene transfer in Crigler Najjar Syndrome. Subjects will receive a single dose of AT342 delivered intravenously. A maximum of 3 dose levels of AT342 are planned for evaluation in this study. Up to four subjects will be enrolled at each dose level including up to 1 subject at each dose level randomized to control with delayed administration of the investigational product. Dose escalation to the next dose level will be considered after evaluation of at least 4 weeks of data from subjects dosed at the current dose level. One of the dose levels will be chosen for dose expansion, and the chosen dose will be administered to all delayed-treatment control subjects.

The primary efficacy endpoint measure of change in total serum bilirubin will be assessed at weeks 12 (whilst still on phototherapy) and week 18 (after phototherapy has been weaned) after administration of AT342; and the primary efficacy endpoint measure of change in number of hours of phototherapy will be assessed at week 18

This study will utilize an independent Data Monitoring Committee that will monitor subject safety and provide recommendations to Audentes regarding dose escalation, dose expansion, and safety matters.

At study termination, only one (1) pediatric participant was enrolled. This study was intended to be a Phase 1/2 trial but the study never moved forward to Phase 2.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has a diagnosis of Crigler-Najjar syndrome resulting from a confirmed mutation in the UGT1A1 gene as assessed by a Sponsor-approved testing facility.
* Subject is aged ≥1 year.
* Subject is prescribed daily phototherapy for a minimum of 6 hours within a 24-hour period (daily illumination time).

Key Exclusion Criteria:

* Subject is currently participating in an interventional study or has received gene or cell therapy.
* Subject has received a whole liver, partial liver, or hepatocyte transplant; or subject has a liver transplant scheduled within the treatment period of this study.
* Subject has significant cholestatic disease at screening.
* Subject is receiving phenobarbital or other known inducer of UGT1A1 within 30 days of screening.
* Subject tests positive for AAV8 neutralizing antibodies with titers above protocol specified threshold.
* Other than as required per protocol, subject has received immune-modulating agents within 3 months before dosing (use of inhaled corticosteroids to manage chronic respiratory conditions is allowed); use of other concomitant medications to manage chronic conditions must have been stable for at least 4 weeks before dosing.
* Subject has any clinically significant laboratory values, in the opinion of the investigator.
* Subject has clinically significant underlying liver disease (other than CN) at screening.
* Subject has a history of, or currently has, a clinically important condition other than CN, in the opinion of the investigator.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (safety and tolerability) | Baseline to Week 24
  Adverse events, serious adverse events, and laboratory abnormalities (including immunological parameters)
Total serum bilirubin | Baseline to Week 12 (on phototherapy) and Baseline to Week 18 (off phototherapy)
  Change in total serum bilirubin
Hours of Phototherapy | Baseline to Week 18
  Change in number of hours of daily phototherapy (daily illumination time)

SECONDARY OUTCOMES:
Phototherapy | Baseline to Week 18
  Proportion of subjects with successful weaning off of phototherapy
UGT Protein | 24 Weeks
  Change in Liver UGT protein expression, DNA, and RNA levels

OTHER OUTCOMES:
Quality of Life Assessment: Pediatric Quality of Life Inventory (PedsQL) | Baseline to Week 18
  Change in quality of life assessment
Caregiver Burden Assessment: Family Impact Module Scores | Baseline to Week 18
  Change in Burden of Disease score
Clinical Global Impression of Severity and of Improvement | Baseline to Week 18
  Change in Investigator assessment of disease severity and improvement

CONTACTS AND LOCATIONS:
Overall Officials: Suyash Prasad, M.D., Study Director — Audentes Therapeutics
Locations (4):
- United States (2):
  - Children's Hospital at Montefiore, The Bronx, New York
  - Clinic for Special Children, Strasburg, Pennsylvania
- Shaare Zedek Medical Center, Jerusalem, Israel
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No